CLINICAL TRIAL: NCT05917704
Title: CAPO: Classical Guitar to Alleviate Parkinson's Disease Symptom Onus
Brief Title: Classical Guitar for Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Christopher Adams, Acting Instructor, University of Washington
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00017748
Record Dates: First submitted 2023-06-06; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; music-based therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guitar then physical therapy (Active Comparator): Subjects will learn classical guitar then have physical therapy sessions.
  Interventions: Other: Guitar then physical therapy
- Physical therapy then guitar (Active Comparator): Subjects will have physical therapy sessions then learn classical guitar
  Interventions: Other: Physical therapy then guitar

INTERVENTIONS:
Other: Guitar then physical therapy — See arm/group descriptions
  Arms: Guitar then physical therapy
Other: Physical therapy then guitar — See arm/group descriptions
  Arms: Physical therapy then guitar

SUMMARY:
The purpose of this study is to understand if training Parkinson's disease patients in classical guitar will improve motor function, mood, and quality of life. While medication has been found to be effective for many Parkinson's disease patients, many patients still have symptoms. Previous studies have found that music and rhythm-based activities can help Parkinson's disease symptoms. A previous study looked at the effect of playing classical guitar on Parkinson's disease symptoms. They found positive changes in Parkinson's disease symptoms that lasted for 6 weeks after the study ended. Further, there were positive changes in depression, anxiety, and quality of life.

DETAILED DESCRIPTION:
Subjects will be asked to take part in classical guitar lessons once a week for six weeks and physical therapy once a week for six weeks. There will be 40 people enrolled in the study. Twenty people will have classical guitar lessons first and physical therapy second. The other twenty people will have physical therapy first and classical guitar lessons second. The study will last a total of 12 weeks. Each session will last 1-2 hours. Sessions will be held at the Northwest Chapter headquarters of the American Parkinson's Disease Association.

Examples of the types of activities subjects will do during the physical therapy sessions include finger exercises, tasks with both hands, tasks while standing, and tasks while walking.

Examples of the types of activities you will do during the classical guitar lessons include playing chords and songs on the guitar.

Subjects will have physical exams and complete questionnaires at the beginning of the study, at six weeks, and at the end of the study.

If subjects have Apple watches, they will be asked to download an application called StrivePD on their watch and iPhone. StrivePD is an application that allows subjects to keep track of their Parkinson's disease symptoms or set medication reminders, for example. When used with an Apple watch, it can automatically record symptoms like tremors. During this study, the StrivePD application will only be used to collect data about what percentage of the day they have tremors and how much they sleep.

ELIGIBILITY:
Inclusion Criteria:

* 50-90 years old
* Diagnosis with Parkinson's disease by a Movement Disorder specialist

Exclusion Criteria:

* Professional musician or formal music training
* Inability to play a classical guitar physically
* Inability to follow instruction
* Receiving physical therapy at the time of the study
* Unable to attend all sessions of study

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-12-12 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in the motor subscore of the Movement Disorder Society Unified Parkinson's Disease Rating Scale Motor Subscale | Baseline, 6 weeks, 12 weeks
  Change in Parkinson's disease rating scale, range 0-32, higher score means more severe Parkinson's disease symptoms

SECONDARY OUTCOMES:
Change in Parkinson's disease Questionnaire-39 | Baseline, 6 weeks, 12 weeks
  Change in scale for quality of life, range 0-100, higher means worse Parkinson's disease symptoms
Change in percent of day with tremor | Baseline, 6 weeks, 12 weeks
  Change in percent of day with tremor from apple watch
Change in Beck Depression Inventory-II | Baseline, 6 weeks, 12 weeks
  depression scale, range 0-63, higher score means worse depression
Change in Apathy evaluation scale total score | Baseline, 6 weeks, 12 weeks
  Change in apathy scale, range 18-72, higher scores means worse apathy
Change in American Parkinson's disease Association symptom tracker score | Baseline, 6 weeks, 12 weeks
  Change in Parkinson's disease symptom tracker, range 0-50, higher scores means worse symptoms
Change in hours of sleep | Baseline, 6 weeks, 12 weeks
  Change in hours of sleep measured from apple watch data

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Adams, MS, MD, Principal Investigator — University of Washington
Locations (1):
- Northwest Chapter of the American Parkinson Disease Association, Seattle, Washington, United States

REFERENCES:
- [Derived] Adams C, Fulton G. A Cross-over Pilot Study on the Effects of Classical Guitar Instruction on Motor and Non-Motor Symptoms in People with Parkinson's Disease. Neurosci Insights. 2025 Mar 24;20:26331055251329878. doi: 10.1177/26331055251329878. eCollection 2025. PMID 40143890